CLINICAL TRIAL: NCT01468168
Title: A Phase II Prospective, Randomized, Double-Masked, Parallel-Group, Multi-centered Study Assessing the Safety and Efficacy of Two Concentrations of DE-101 Ophthalmic Suspension Compared to Placebo for the Treatment of Dry Eye Disease
Brief Title: A Study Assessing the Safety and Efficacy of DE-101 Ophthalmic Suspension in Dry Eye Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 26-005
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- DE-101 Ophthalmic Suspension High Dose (Experimental)
  Interventions: Drug: DE-101 Ophthalmic Suspension
- DE-101 Ophthalmic Suspension Low Dose (Experimental)
  Interventions: Drug: DE-101 Ophthalmic Suspension
- DE-101 Ophthalmic Suspension Vehicle (Placebo Comparator)
  Interventions: Drug: DE-101 Ophthalmic Suspension Vehicle

INTERVENTIONS:
Drug: DE-101 Ophthalmic Suspension — Ophthalmic suspension; QID
  Arms: DE-101 Ophthalmic Suspension High Dose
Drug: DE-101 Ophthalmic Suspension — Ophthalmic suspension; QID
  Arms: DE-101 Ophthalmic Suspension Low Dose
Drug: DE-101 Ophthalmic Suspension Vehicle — Ophthalmic suspension vehicle; QID
  Arms: DE-101 Ophthalmic Suspension Vehicle

SUMMARY:
To investigate the safety and efficacy of DE-101 to improve the signs and symptoms in dry-eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals considered for entry into the study will be of either sex and any race who have:
* a confirmed diagnosis of dry eye,
* are willing to use no ocular treatments during the study other than study medication,
* have a corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity score of +0.7 logarithm of the minimum angle of resolution (logMAR) or better in each eye,
* will not use contact lenses during the study,
* Females of child-bearing potential must have a negative urine pregnancy test and be willing to use an acceptable method of contraception to be eligible for, and continue participation in, the study,
* 18 years of age or older,
* able to understand and provide written informed consent

Exclusion Criteria:

* Subjects with any of the following are not eligible to participate in the study:
* Fluorescein corneal staining or conjunctival staining that is too severe
* Conditions requiring the use of ophthalmic prescription or over the counter medications during the study (except for study medications)
* Any type of current punctal occlusion including punctal plugs, intracanalicular punctal plugs or cauterized puncta
* Any type of ocular surgery within 90 days prior to Visit 1 (Day 1)
* Known history of Steven-Johnson's syndrome, Riley-Day syndrome, and/or ocular pemphigoid
* Ocular(including lid)disease/abnormality that may interfere with the study
* Corneal transplant in either eye, at any time prior to enrollment in the study
* Laser refractive surgery less than one year prior to Visit 1 (Day 1)
* Conditions requiring the use of any systemic medication that is not ongoing at a stable dosage for at least 30 days prior to Visit 1 (Day 1)
* Application of isotretinoin within 30 days prior to Visit 1 (Day 1)
* Known allergy or sensitivity to any of the study medication components
* Uncontrolled systemic conditions or other conditions which would confound the study evaluations or endanger the safety of the subject
* A woman who is pregnant, nursing, or planning a pregnancy
* Participation in another investigational drug or vaccine trial, or participation in such a trial within 30 days prior to Visit 1 (Day 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Tear volume increase from baseline | baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - New Port Beach, California
  - Parker, Colorado
  - Largo, Florida
  - Morrow, Georgia
  - Roswell, Georgia
  - Bangor, Maine
  - Kansas City, Missouri
  - St Louis, Missouri
  - Washington, Missouri
  - High Point, North Carolina
  - Cleveland, Ohio
  - Salt Lake City, Utah
  - Norfolk, Virginia